CLINICAL TRIAL: NCT04551261
Title: A Phase I, Single-center, Open Label Clinical Study, to Evaluate the Pharmacokinetic Character of GLS4 Combined With RTV or TAF Alone or GLS4 and RTV and TAF Combination Administration in Healthy Subjects
Brief Title: GLS4/RTV and TAF Drug-drug Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PCD-DGLS4-20-001
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2021-05

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ritonavir; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Subjects will receive GLS4 and RTV on Day 1, TAF on Day 5-14, GLS4 and RTV and TAF on Day15.
  Interventions: Drug: GLS4; Drug: RTV; Drug: TAF
- Part B (Experimental): Subjects will receive TAF on Day 1, GLS4 and RTV on Day 5-14, GLS4 and RTV and TAF on Day15.
  Interventions: Drug: GLS4; Drug: RTV; Drug: TAF

INTERVENTIONS:
Drug: GLS4 — It is a new dihydropyrimidine antiviral drug that interferes the assembly of HBV core granule.
Drug: RTV — 1. It is HIV protease inhibitors indicated in combination with other antiretroviral agents for the treatment of HIV-1 infection;
  2. It is a CYP3A inhibitor combined with other drug to increase the exposure in human.
  Other Names: ritonavir
Drug: TAF — It is a hepatitis B virus (HBV) nucleoside analog reverse transcriptase inhibitor and is indicated for the treatment of chronic hepatitis B virus infection in adults with compensated liver disease.
  Other Names: tenofovir alafenamide

SUMMARY:
The purpose of this study is to evaluate the drug-drug-interaction (DDI), pharmacokinetics (PK) and tolerability of GLS4/RTV combined with TAF in healthy subjects.

DETAILED DESCRIPTION:
This is a 2-part study with each part is an open-label study in healthy adult subjects.

Total 28 subjects will be enrolled into the study and divided into 2 part (Part A and Part B), 14 subjects in each part. With each part, the subject will be receive study drug per the defined treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 50 years of age, inclusive, at Screening;
* Body mass index between 18.0 and 28.0 kg/m2, inclusive, at Screening;
* Females of childbearing potential and male subjects will agree to use contraception from screening to the 6 months after the last administration.

Exclusion Criteria:

* In the 12 months prior to screening, observing clinical significance of the following diseases, including but not limited to, gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental, or cardio-cerebrovascular diseases;
* Allergic constitution (multiple drug and food allergies);
* A history of alcoholism;
* Take any prescription drug, over-the-counter drug, vitamin product or herbal medicine within 14 days of screening;
* Any drug that changes the liver enzyme activity, such as barbiturates and Rifampicin, was taken within 30 days before screening;
* P-GP, BCRP, OATP1B1, OATP1B3, OAT1, OAT3 or MRP4 inhibitors or inducers, such as azithromycin, pantoprazole or St. John's herb, etc., was taken within 30 days before screening;
* Female subjects are lactating or have positive blood pregnancy results during the screening period;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Cmax | predose to 96 hour after dosing
  maximum observed plasma concentration
AUC | predose to 96 hour after dosing
  area under the plasma concentration-time curve (AUC)
Adverse event | Baseline to day 22
  To assess the safety and tolerability of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No